CLINICAL TRIAL: NCT06609083
Title: Effect of Cannabinoids on Tobacco Product Demand and Pharmacodynamics: Cigarette Use
Brief Title: Effect of Cannabis on Cigarette Use Behavior
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: IRB00435111; R01DA058624 (NIH)
Record Dates: First submitted 2024-09-20; First posted 2024-09-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Cannabis Use; Tobacco Use; Cigarette Smoking
Keywords: cannabis; cigarette; marijuana; THC; tobacco
MeSH Terms: conditions — Tobacco Use; Cigarette Smoking; Marijuana Abuse | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Smoked THC (Experimental): Each participant in this arm will receive 0, 5, and 30mg of THC over the course of six visits. Each participant will also receive combustible cigarettes containing 0.03mg and 0.80mg of nicotine.
  Interventions: Drug: THC 30mg; Drug: THC 5mg; Drug: THC 0mg; Drug: Cigarette Full Nicotine; Drug: Cigarette Reduced Nicotine
- Vaporized THC (Experimental): Each participant in this arm will receive 0, 5, and 30mg of THC over the course of six visits. Each participant will also receive combustible cigarettes containing 0.03mg and 0.80mg of nicotine.
  Interventions: Drug: THC 30mg; Drug: THC 5mg; Drug: THC 0mg; Drug: Cigarette Full Nicotine; Drug: Cigarette Reduced Nicotine

INTERVENTIONS:
Drug: THC 30mg — High dose of THC (30 mg)
Drug: THC 5mg — Low dose of THC (5 mg)
Drug: THC 0mg — Placebo dose of THC (0 mg)
Drug: Cigarette Full Nicotine — Full nicotine cigarette
Drug: Cigarette Reduced Nicotine — Reduced nicotine cigarette

SUMMARY:
The purpose of this study is to determine the impact of tetrahydrocannabinol (THC) administration on motivational, subjective, and physiological effects of cigarettes. The study's goals are to test demand for cigarettes, tobacco craving, affect, heart rate, blood pressure, expired breath carbon monoxide, and cognitive performance. Researchers will compare multiple doses of THC and a placebo in participants who smoke cigarettes and either smoke or vape THC in the laboratory.

DETAILED DESCRIPTION:
A full-factorial laboratory study will be conducted to determine the impact of acute THC administration on the dose-related motivational, subjective, and physiological effects of combustible cigarettes. This study will employ a double-blind, placebo-controlled, within-subjects crossover design to examine the dose-effects of THC on combustible tobacco use. The study will use multiple active doses of THC and placebo (0, 5, and 30 mg; corresponding to 0, 1, and 6 standard THC unit doses). Participants will be randomized to either smoked or vaporized THC administration using a between-subjects approach to evaluate the effect of congruent versus incongruent routes of THC and tobacco administration on study outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy non-treatment seeking adults aged 21 or older
2. Report daily use of combustible tobacco cigarettes
3. Biological confirmation of cigarette use: have an expired carbon monoxide (CO) level of more than 5 ppm and a positive urine cotinine test at screening
4. Report current use of cannabis (at least 1 occasion per week)
5. Have experience with the inhalation route of administration for cannabis
6. Biological confirmation of cannabis use: have a positive urinary THC drug test at screening.
7. For women of children bearing potential and men with female partners of child-bearing potential, must be willing to use an effective form of contraception during the study.

Exclusion Criteria:

1. Report current intention to reduce or quit cannabis or tobacco use within the next 30 days
2. Meet Diagnostic and Statistical Manual (DSM-5) criteria for a substance use disorder other than alcohol, cannabis, or nicotine
3. Test positive for illicit drugs other than cannabis and tobacco
4. Positive breath alcohol test at study admission
5. Have a current physical or mental illness judged by the study team to negatively impact participant safety or scientific integrity
6. Have a lifetime history of suicidal behavior (i.e. past suicide attempt), or current suicidal behavior or ideation as assessed by the Columbia Suicide Severity Rating Scale (C-SSRS)
7. Are currently pregnant, planning to become pregnant in the next three months or are currently breastfeeding
8. Have a history of clinically significant cardiac arrhythmias or vasospastic disease (e.g., Prinzmetal's angina)
9. Are currently enrolled in another clinical trial or have received any drug as part of a research study within 30 days of study participation.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2029-04-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Demand Intensity | 45 minutes after THC or placebo administration
  Consumption of cigarette puffs at unconstrained price as measured by an incentivized demand task. Minimum value is 0, maximum value is not constrained. Higher scores indicate more consumption at unconstrained price (a worse outcome).
Demand Elasticity | 45 minutes after THC or placebo administration
  Changes in cigarette consumption with changes in price as measured by an incentivized demand task. There is no minimum or maximum value. Higher scores indicate greater cigarette price sensitivity (a better outcome).

SECONDARY OUTCOMES:
Minnesota Nicotine Withdrawal Scale (MNWS) | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  A subjective effect measure of nicotine withdrawal. Minimum value is 0, maximum value is 68. Higher scores indicate greater nicotine withdrawal (a worse outcome). Primary outcomes will be the peak change from baseline.
Brief Questionnaire of Smoking Urges (QSU - Brief) Factor 1 | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  Self report assessment smoking urges. Factor 1 - Intention/Desire to Smoke. Score minimum is 7, Score Maximum is 35. Primary outcomes will be the peak change from baseline.
Brief Questionnaire of Smoking Urges (QSU - Brief) Factor 2 | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  Self report assessment smoking urges. Factor 2 - Relief of Negative Affect & Urgent Desire to Smoke. Score minimum is 7, Score Maximum is 35. Primary outcomes will be the peak change from baseline.
Drug Effect Questionnaire for Like Drug | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  The Drug Effect Questionnaire will be administered using a visual analog scale. Participants place a mark on a 100mm line with the left endpoint labeled Not at All and the right endpoint labeled Extremely. Primary outcomes will be the peak change from baseline.
Heart Rate | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  Heart rate will be recorded using an automated vital signs monitor to monitor safety and provide an objective index of the time course and magnitude of drug effects. Primary outcomes will be the peak change from baseline.
Diastolic Blood Pressure | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  Diastolic Blood Pressure will be recorded using an automated vital signs monitor to monitor safety and provide an objective index of the time course and magnitude of drug effects. Primary outcomes will be the peak change from baseline.
Systolic Blood Pressure | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  Systolic Blood Pressure will be recorded using an automated vital signs monitor to monitor safety and provide an objective index of the time course and magnitude of drug effects. Primary outcomes will be the peak change from baseline.
Divided Attention Task (DAT) Performance | Baseline, 15 minutes, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, and 6 hours post THC or placebo administration.
  Participants will complete a Divided Attention Task (DAT) in which the participant must simultaneously track a stimulus moving horizontally on a computer screen and respond to visual stimuli presented. The primary dependent measure is the average distance maintained from the target stimulus. Primary outcomes will be the peak change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Dustin Lee, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University Behavioral Pharmacology Research Unit, Baltimore, Maryland, United States